CLINICAL TRIAL: NCT04245280
Title: Effectiveness of Pericapsular Nerve Group (PENG) Block Combined to Lateral Femoral Cutaneous Nerve (LFCN) Block on the Quality of Recovery After Total Hip Replacement
Brief Title: Effectiveness of PENG Block Combined to LFCN Block on the Quality of Recovery After Total Hip Replacement
Acronym: PENG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19.275
Record Dates: First submitted 2020-01-22; First posted 2020-01-28 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Total Hip Replacement Surgery; Postoperative Pain
Keywords: Regional anesthesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Prospective, randomized controlled, triple blind
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: triple blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG and LFCN blocks with ropivacaine (Active Comparator): For the PENG block, and after negative aspiration, 20 ml of a solution of ropivacaine 0.5% with epinephrine 2.5 mcg/ml will be injected in 5 ml aliquots. Then, for the LFCN block, the lateral femoral cutaneous nerve will be localized, infero-medially to the antero-superior iliac spine, superficially to the sartorius muscle and 5 ml of the same solution will be injected with the same needle.
  Interventions: Drug: Ropivacaine 0.5% Injectable Solution
- PENG and LFCN blocks with saline solution (Placebo Comparator): For the PENG block, and after negative aspiration, 20 ml of a saline solution will be injected in 5 ml aliquots. Then, for the LFCN block, the lateral femoral cutaneous nerve will be localized, infero-medially to the antero-superior iliac spine, superficially to the sartorius muscle and 5 ml of the same saline solution will be injected with the same needle.
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Ropivacaine 0.5% Injectable Solution — ropivacaine 0.5% with epinephrine 2.5 mcg/ml
  Other Names: Ropivacaine 0.5%
  Arms: PENG and LFCN blocks with ropivacaine
Drug: Saline Solution — normal saline solution (NaCl 0.9%)
  Other Names: Placebo
  Arms: PENG and LFCN blocks with saline solution

SUMMARY:
The main objective of this study is to evaluate the effectiveness of the association of PENG and LFCN blocks on the quality of recovery 24 hours after total hip replacement surgery.

DETAILED DESCRIPTION:
Total hip replacement is a frequent procedure in the geriatric population associated with moderate post-operative pain. It is known that a sub-optimal analgesia is associated with a delayed mobilization leading to a longer hospital stay, poor functional recovery and increased thromboembolic complications. Moreover, opioid analgesia, especially in the geriatric population, increases the incidence of delirium.

Multimodal analgesia, combining different analgesic classes and regional anesthesia, is preferable than relying mainly on opioids, improving the outcomes in the post-operative period. Until now, no regional anesthesia technique has proven itself to be better than the others, each having its limitations. While the local anesthetic doses are high with the peri-articular infiltration under direct visualisation, the epidural is associated with bilateral block and sympathetic block. Also, the lumbar plexus block is a technically difficult block and is associated with a motor block. Finally, other blocks such as the femoral, 3:1 or fascia iliaca are not blocking the totality of the nerves involved in the post-operative pain pathways.

A recent anatomic study from Short et al. demonstrated a greater implication than what was previously known of the accessory obturator nerve and the femoral nerve in the etiology of the post-operative pain. Regarding the incision, it is generally located in the lateral femoral cutaneous nerve territory. Recently published as case reports, the PENG block is a new regional anesthesia technique that has emerged for hip surgeries. It consists of injecting local anesthetics in the myofascial plan between the psoas anteriorly and the pubic ramus posteriorly.

With this prospective randomized trial, the investigators aim to investigate whether a PENG block combined with the LFCN block provides a superior analgesia compared to multimodal analgesia alone and improves the outcomes of the patients in the post-operative phase.

Methods:

The PENG and LFCN blocks will be performed with the patients in a dorsal decubitus position, using a high frequency linear ultrasound probe (Sonosite HFL50 6-15 MHz) in the inguinal area, with an insulated hyperechoic needle (50-80 mm, 22 gauge, Pajunk) placed in plane in relation to the ultrasound beam. The myofascial plane between the psoas anteriorly and the pubic ramus posteriorly will be targeted. The anesthesiologist will confirm the correct position of the needle by injecting 1 ml of 5% dextrose.

For the group A, after negative aspiration, 20 ml of a solution of ropivacaine 0,5% with epinephrine 2,5 mcg/ml will be injected in 5 ml aliquots. Then, the lateral femoral cutaneous nerve will be localized, infero-medially to the antero-superior iliac spine, superficially to the sartorius muscle and 5 ml of the same solution will be injected with the same needle. For group B, the technique of the blocks will be identical to group A, but 20 ml and 5 ml of a sterile saline solution will be used instead.

Patients will then be taken to the operating room where a spinal anesthesia will be performed using 12 mg of iso or hyperbaric bupivacaine (at the discretion of the anesthesiologist) with the addition of 15 mcg of fentanyl. A dose of 8 mg of dexamethasone will be administered intravenously over 10 minutes. In case of failed spinal anesthesia, patient will be excluded from the study.

For hospitalized patients:

In the absence of contraindication, patient controlled analgesia (PCA) with hydromorphone will be prescribed post-operatively, until 8h on post-operative day 1. Patients will thus have the possibility to self-administer 0,2 mg of hydromorphone every 5 minutes, for a maximum of 10 doses per hour. In case of contraindications, subcutaneous or per os hydromorphone will be prescribed to these patients. Multimodal analgesia with acetaminophen and celecoxib (in absence of contraindication) will be continued as per protocol.

For patients treated on an outpatient trajectory:

Patients will benefit from medical prescriptions for total hip replacement, including hydromorphone or oxycodone, celecoxib and acetaminophen.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old undergoing a total hip replacement surgery

Exclusion Criteria:

* Contraindication to regional anesthesia (allergy to local anesthetics, severe coagulopathy, infection in the designated area, pre-existing neuropathy in the obturator or femoral territory)
* Contraindication to spinal anesthesia
* Patient's refusal or inability to consent
* Opioid use on a regular basis pre-operatively
* Inability to communicate with medical team or research team
* Inability to understand the items of the multiple forms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Quality of recovery, QoR15 (Quality of Recovery 15) | Change between baseline (day 0) and post-operative day 1
  QoR15 is a valid questionnaire to measure the quality of recovery after surgery and anaesthesia, which includes 15 questions. Each of the 15 items are scored by the patient from 0 (worst score) to 10 (optimal score), giving a lowest possible score of 0 (worst outcome), and a highest possible score of 150 (optimal outcome).

SECONDARY OUTCOMES:
Verbal numeric rating scale (vNRS) for pain assessment | 8 hours, 16 hours and 24 hours after the surgery
  Postoperative pain assessment will be performed using the vNRS; score (0 = no pain, 10 = unbearable pain). The vNRS scores at rest and after mobilisation (15° hip flexion) will be recorded at postoperative 8, 16 and 24 hours.
Difficulty of realization of the block | At the end of the blocks on Day 0
  Numeric scale from 1 to 5 describing the difficulty of the block based on a local scale that has not been validated. (Score 1= Easy site identification, good needle positioning and adequate dispersion of the solution on the first try; Score 2= Difficulty in identifying the site but positioning and dispersion of the solution on the first try once it has been identified; Score 3= one repositioning of the needle necessary, adequate dispersion thereafter; Score 4= More than one repositioning necessary, adequate dispersion thereafter; Score 5= Dispersion remains suboptimal despite several repositionings of the needle.
Mild cognitive impairment assessment using the Montreal Cognitive Assessment (MoCA) | Pre-operative day 0 (day before or morning of the surgery) and Post-operative day 1
  The incidence of mild cognitive impairment in patients will be evaluated using the MoCA screening validated tool (Score 0-30; higher score indicates better performance) for hospitalized patients.
  For patients with an outpatient trajectory, the incidence of mild cognitive impairment in patients will be evaluated using the MoCA BLIND screening validated tool (Score 0-22; higher score indicates better performance). Then the 22-point telephone MoCA will be converted to 30 points for comparison purposes as proposed by Katz et al. 2021
Opioids side effects | 8 hours, 16 hours and 24 hours after the surgery
  The presence or absence of opioids side effects such as drowsiness, desaturation (only for hospitalized patients), nausea and vomiting will be recorded over a 24 hours period after the surgery.
Quadriceps weakness | On post-operative day 1
  Presence of weakness of the quadriceps using a scale where 0= no effect; 1 = knee flexion possible but not hip flexion; 2 = absence of knee and hip flexion.
In-hospital stay for hospitalized patients | An average of 1 to 2 days
  Number of days of hospital stay for patients.
Walking distance after the surgery for hospitalized patients | On post-operative day 1
  The walking distance accompanied by a physiotherapist will be recorded.
Number of participants with block complications | On post-operative day 1
  Any complications or side effects of the blocks will be recorded and addressed to insure the safety of the patients, such as local infection, intravascular injection of local anesthetics and immediate systemic toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Garneau, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No